CLINICAL TRIAL: NCT02633254
Title: Targeted Vessel Ablation of Type 3 Uterine Fibroids With Magnetic Resonance Guided High Intensity Focused Ultrasound
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Maurice A.A.J. van den Bosch, Prof. Dr., UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-528
Record Dates: First submitted 2015-11-19; First posted 2015-12-17 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Uterine Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): Treatment group Magentic Resonance guided High Intensity Focused Ultrasound will be employed on uterine fibroids
  Interventions: Device: Magnetic Resonance guided High Intensity Focused Ultrasound

INTERVENTIONS:
Device: Magnetic Resonance guided High Intensity Focused Ultrasound — Targeted vessel ablation of type 3 uterine fibroids with magnetic resonance guided high intensity focused ultrasound

SUMMARY:
So-called type 1 and 2 uterine fibroids are well treatable with Magnetic Resonance guided High Intensity Focused Ultrasound (MR-HIFU). The other type, type 3 fibroids, however, are known for their high perfusion and poor treatment outcome after MR-HIFU. This study proposes a new strategy to treat type 3 fibroids with MR-HIFU. Very precise, small, high-power sonications (heating points) will be used to occlude (part of) the feeding vessels of the fibroid. This deminishes the negative effect of the high perfusion and is hypothesized to transform a type 3 fibroid into a type 2 or possibly even a type 1 fibroid. Consequently, the bulk volume of the fibroid can be treated using the standard approach.

DETAILED DESCRIPTION:
Rationale: Uterine fibroids or leiomyomas are common benign tumors that arise from smooth muscle cells of the uterus with a prevalence ranging from 20% to 40% in reproductive aged women. Invasive treatments, such as hysterectomy and myomectomy, represent the golden standard with respect to therapy. Alternatively, uterine artery embolization is offered as a less invasive option. However, to date the only non-invasive technique is high intensity focused ultrasound (HIFU) ablation. HIFU ablation uses focused ultrasound waves to non-invasively heat and thermally ablate tissue. Combined with magnetic resonance guidance (MR-HIFU) this allows an entirely non-invasive intervention with anatomical 3D images for the planning of the treatment volume, and real-time temperature monitoring for therapeutic guidance.

A limitation of MR-HIFU is that currently not all types of uterine fibroids are treatable. With respect to MR-HIFU treatment, uterine fibroids are classified in three classes based on the signal intensity of T2-weighted MR images. While MR-HIFU has been shown to result in a reliable positive therapeutic outcome in type 1 and type 2 fibroids, the therapeutic success in type 3 fibroids has so far been limited. The current clinical consensus is that the high perfusion in type 3 fibroids, which causes the heat deposited by the HIFU to be rapidly evacuated from the treatment site, results in insufficient temperatures to induce necrosis in the fibroids. Therefore, a new treatment strategy is proposed to effectively treat type 3 fibroids with MR-HIFU.

Objective: To investigate whether it is possible to manipulate perfusion in type 3 fibroids with MR-HIFU.

Study design: Single-center, single arm, non-randomized trial. Ten patients will be treated.

Study population: Adult women with a type 3 uterine fibroid who fulfill the in- and exclusion criteria.

Intervention: During the MR-HIFU treatment, the local vascular feeding network will be selectively targeted first with high power sonications with the intention to reduce or interrupt the perfusion of the entire fibroid volume. Subsequently, the remaining fibroid volume will be ablated, similar to the treatment approach of type 1/2 fibroids.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The fibroid type and the eligibility for MR-HIFU treatment will be determined on a clinically obtained MRI scan. The results of the scan and information about this study are provided to the patient during a phone call. If the patient is interested, the study information is sent by mail. The patient receives a second phone call to ask if she wishes to participate. If so, an appointment at the hospital is arranged to give details on the study, answer questions, and show the clinical MR scan. If the patient still wants to participate, informed consent (IC) is signed. The HIFU treatment will be scheduled in consultation with the patient.

Patients will be sedated during the HIFU intervention, as it is also the case during the standard HIFU treatment of type 1/2 fibroids. Compared to the standard HIFU treatment, the initial selective ablation of the vascular feeding network with high power sonications will be added. The subsequent therapy for the remainder of the fibroid will follow the standard therapeutic HIFU treatment of type 1/2 fibroids.

One week after the treatment the patient will receive a phone call to ask about adverse events. Three months after the treatment a follow-up MR scan, including a DCE scan, will be performed. In addition, the patient will be asked about any adverse events that might have occurred during a phone call.

Potential adverse effects include skin burns due to heating of the cutaneous and sub-cutaneous abdominal fat and risk of abdominal pain due to the occlusion of the vascular network. To mitigate the risk of skin burns, a cooling cushion is integrated in the HIFU table top and will protect the skin and part of the abdominal fat from overheating.

If women with a type 3 fibroid do not want to participate in this study, they are not eligible for MR-HIFU treatment and are referred by their gynecologist to a more invasive treatment option like uterine artery embolization or hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent;
* A type 3 uterine fibroid;
* Sufficient physical condition to undergo deep sedation;
* Waist circumference that allows positioning on the HIFU table top inside the MR bore.

Exclusion Criteria:

* Contra-indication for MRI scanning according to the hospital guidelines;
* Contra-indication to injection of gadolinium-based contrast agent, including known prior allergic reaction to any contrast agent, and renal failure (GFR <30 mL/min/1.73 m2);
* Surgical clips or considerable scar tissue in the HIFU beam path;
* A total of more than ten fibroids;
* Post- or peri-menopausal status;
* Fibroid size >10 cm in diameter;
* Patient has an active pelvic infection;
* Patient has an undiagnosed pelvic mass outside the uterus;
* Patient who is not able to tolerate the required stationary prone position during treatment.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Time to peak | three months
  The main endpoint of this feasibility study is the manipulation of perfusion in the type 3 uterine fibroid. The perfusion will be assessed by comparing the results of dynamic contrast-enhanced MRI (DCE-MRI) before and after treatment and after three months, i.e. the time to peak values. Data will be analyzed using Philips IntelliSpace Portal.
Regional Blood volume | Three months
  The main endpoint of this feasibility study is the manipulation of perfusion in the type 3 uterine fibroid and the possibly related adverse events. The perfusion will be assessed by comparing the results of dynamic contrast-enhanced MRI (DCE-MRI) before and after treatment and after three months, i.e. regional blood volumes (area under the curve). Data will be analyzed using Philips IntelliSpace Portal.

SECONDARY OUTCOMES:
Adverse effects | Three months
  The adverse events will be reported in the case report form (CRF) based on the assessments one week and three months post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Maurice van den Bosch, Prof Dr, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No